CLINICAL TRIAL: NCT00706199
Title: Analysis of Expression of Antigens in Bone Marrow Samples From Volunteering Donors.
Brief Title: The Expression of Antigens in Bone Marrow Samples From Volunteering Donors.
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111684
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Cancer
Keywords: bone marrow; antigen expression; volunteers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group A: donors
  Interventions: Procedure: Bone marrow aspiration

INTERVENTIONS:
Procedure: Bone marrow aspiration — Collection of a 2 ml bone marrow sample from an aspirate carried out for medical purposes.

SUMMARY:
Antigen expression levels in bone marrow from volunteering donors will be analyzed. The results of this analysis will be used to establish a clinical test to identify cancer patients who could qualify to receive an investigational treatment being developed by GlaxoSmithKline.

ELIGIBILITY:
Inclusion Criteria:

* The donor is aged >= 18 years
* Written informed consent has been obtained prior to the performance of any specific procedure.
* The donor has a medical indication for which a bone marrow aspiration is planned.
* The donor is eligible for a bone marrow aspiration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-07-03; Primary Completion 2009-01-23 (Actual); Study Completion 2009-01-23 (Actual)

PRIMARY OUTCOMES:
Number of copies of Wilms' Tumor 1 (WT1) antigen expression in bone marrow | At Day 0
  Establishment of the range of WT1 transcript levels in a collection of bone marrow samples by real-time quantitative RT-PCR (Reverse Transcription Polymerase Chain Reaction). Due to the low numbers, they were expressed as [value x 10E-03]. Only the samples with gene expression >0 were presented.
Number of copies of PRAME (Preferentially expressed in melanoma)antigen expression in bone marrow | At Day 0
  Establishment of the range of PRAME transcript levels in a collection of bone marrow samples by real-time quantitative RT-PCR (Reverse Transcription Polymerase Chain Reaction). Due to the low numbers, they were expressed as [value x 10E-03]. Only the samples with gene expression >0 were presented.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ottignies, Belgium